CLINICAL TRIAL: NCT05546255
Title: Phase II Clinical Study of Eribulin Mesylate Combined With Lobaplatin in the Treatment of Recurrent or Metastatic Triple-negative Breast Cancer
Brief Title: Eribulin Mesylate Combined With Lobaplatin in the Treatment of Recurrent or Metastatic Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-006461
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin; lobaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin Combined With Lobaplatin (Experimental): Eribulin 1.4mg/m2 d1 Lobaplatin 25g/m2 d1 / q14d
  Interventions: Drug: Eribulin Mesylate; Drug: Lobaplatin

INTERVENTIONS:
Drug: Eribulin Mesylate — The recommended dose of Eribulin is 1.4 mg/m2 administered intravenously over 2 to 5 minutes on Days 1
Drug: Lobaplatin — The recommended dose of lobaplatin is 25mg/m2 administered intravenously over on Days 1

SUMMARY:
A prospective phase II study conducted at the Cancer Hospital Chinese Academy of Medical Sciences to compare the effectiveness of eribulin combined with lobaplatin in the treatment of recurrent or metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
This study is designed to be a prospective phase II study conducted at the Cancer Hospital Chinese Academy of Medical Sciences. The target populations of this study are patients with recurrent or metastatic triple-negative breast cancer who received the therapy of eribulin combined with lobaplatin from July 1, 2020 to December 31, 2022. It is expected to enroll 40 subjects in this study. The subjects' data such as demographics and other baseline characteristics, medications, prognosis, will be collected, and statistical analysis of data will be conducted to compare the effectiveness outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 18 and 75
2. Recurrence or metastasis OF TNBC confirmed by histological or cytological methods, TNBC definitions of ER, PR and HER-2 are negative, if there is metastasis pathology, the histological pathology of metastasis shall prevail.ER and PR negative were defined as ER < 10% positive and PR < 10% positive.
3. Disease progression after at least one prior systemic treatment and anthracycline and/or taxane use;Note: For neoadjuvant/adjuvant therapy, recurrence or disease progression during treatment or within 6 months of discontinuation of treatment should be counted as first-line systemic treatment failure;
4. There should be at least one measurable lesion according to the efficacy evaluation criteria for solid tumors (RECIST version 1.1)

Exclusion Criteria:

1. The number of previous treatment lines (including postoperative adjuvant therapy) <2 lines
2. symptomatic central system metastases. Patients with stable asymptomatic BMS who have received brain radiation and who have at least one other evaluable target in addition to the BMS can be enrolled (evaluable target should be at least 4 weeks away from the last radiotherapy).
3. New bisphosphonate or dinoselmer treatment for bone metastases was initiated within 28 days prior to study initiation.(Subjects are permitted if they have already been treated with bisphosphonate or dinoselmer for at least 4 weeks of optimal stable administration prior to study initiation.)Subjects already enrolled in this study may begin treatment with bisphosphonate or dinoselmer for bone metastases after the first post-treatment evaluation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 1 year after the last patient enrolled
  ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival | up to 1 year after the last patient enrolled
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause
adverse events | approximately 1.5 years
  Incidence and Severity of adverse events, such as hematologic, hepatotoxicity，Incidence of hypertension，Incidence of proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China